CLINICAL TRIAL: NCT03290950
Title: Daratumumab, Carfilzomib, Lenalidomide, and Dexamethasone in Newly-Diagnosed Multiple Myeloma: A Clinical and Correlative Phase II Study
Brief Title: A Study of Daratumumab in Patients With Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-352
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Daratumumab; Carfilzomib; Lenalidomide; Dexamethasone; 17-352
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Phase II study and treated with 4-drug combination of daratumumab, carfilzomib, lenalidomide, and dexamethasone.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Single arm, two-stage phase II trial of combination therapy (daratumumab, carfilzomib, lenalidomide, and dexamethasone for newly diagnosed multiple myeloma patients. Patients achieving ≥PR at end of 4 cycles will continue to receive the planned total of 8 cycles of combination therapy. Patients may go onto receiving additional maintenance phase therapy with lenalidomide under a separate treatment protocol. Patients ≤ PR after completing 4 cycles will go off study therapy.
  Interventions: Drug: daratumumab; Drug: carfilzomib; Drug: lenalidomide; Drug: dexamethasone
- Cohort 2 (Experimental): Single arm, two-stage phase II trial of combination therapy (daratumumab, carfilzomib, lenalidomide, and dexamethasone for newly diagnosed multiple myeloma patients. Patients achieving ≥PR at end of 4 cycles will continue to receive the planned total of 8 cycles of combination therapy. Patients may go onto receiving additional maintenance phase therapy with lenalidomide under a separate treatment protocol. Patients ≤ PR after completing 4 cycles will go off study therapy.
  Interventions: Drug: daratumumab; Drug: carfilzomib; Drug: lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: daratumumab — Cycle 1 ONLY: Daratumumab 16 mg/kg days 1, 8, 15, and 22, Cycle 2: Daratumumab 16mg/kg days 1, 8, 15, and 22; Cycles 3-6: Daratumumab 16mg/kg days 1 and 15, Cycles 7-8: Daratumumab 16mg/kg day 1; Daratumumab rate of infusion is per MSKCC guidelines.
Drug: carfilzomib — Cycle 1 ONLY: Carfilzomib 20 mg/m2 per dose, days 2 and 3; Carfilzomib 36 mg/m2 per dose, days 8, 9, 15, and 16; Cycles 2-8: Carfilzomib 36 mg/m2 per dose, days 1, 2, 8, 9, 15, and 16
Drug: lenalidomide — Cycle 1 ONLY: Lenalidomide 25 mg/day, days 2-21 every 28 days; Cycles 2-8: Lenalidomide 25 mg/day, days 1-21 every 28 days
Drug: dexamethasone — Cycle 1 ONLY: Dexamethasone 20 mg/dose, days 2, 3, 8, 9, 15, 16, Cycles 2: Dexamethasone 20mg/dose, days 1, 2, 8, 9, 15, 16 and 22; Cycles 3-4: Dexamethasone 20mg/dose, days 1,2,8,9,15 and 16, Cycles 5- 8: Dexamethasone 10mg/dose, days 1, 2, 8, 9, 15, and 16
  Other Names: Cohort 1 administration
  Arms: Cohort 1
Drug: dexamethasone — Cycle 1 ONLY: Dexamethasone 20 mg/dose, days 1, 2, 22; 40 mg/dose days 8 and 15, Cycles 2: Dexamethasone 40mg/dose, days 1, 8, 15; 20 mg/dose day 22, Cycles 3-4: Dexamethasone 40mg/dose, Days 1, 8 15, Cycles 5-8: Dexamethasone 20mg/dose, Days 1, 8, 15
  Other Names: Cohort 2 administration
  Arms: Cohort 2

SUMMARY:
This is a study to test the safety and effectiveness of the study drug, daratumumab in combination with carfilzomib, lenalidomide and dexamethasone. The purpose of this study is to test whether giving daratumumab along with the other drugs (carfilzomib, lenalidomide and dexamethasone) is safe for patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with histologically confirmed MM based on the following criteria:

  * Clonal plasma cells in the bone marrow
  * Measurable disease within the past 4 weeks defined by any one of the following:
  * Serum monoclonal protein ≥ 1.0 g/dL
  * Urine monoclonal protein >200 mg/24 hour
  * Involved serum immunoglobulin free light chain > 10 mg/dL AND abnormal kappa/lambda ratio
* Evidence of underlying end organ damage and/or myeloma defining event attributed to underlying plasma cell proliferative disorder meeting at least one of the following:

  * Hypercalcemia: serum calcium >0.25 mmol/L (> 1 mg/dL) above upper limit of normal or ≥ 2.75 mmol/L (11 mg/dL)
  * Anemia: hemoglobin value <10 g/dL or > 2 g/dL below lower limit of normal
  * Bone disease: ≥ 1 lytic lesions on skeletal X-ray, CT, or PET-CT. For patients with 1 lytic lesion, bone marrow should demonstrate ≥10% clonal plasma cells
  * Clonal bone marrow plasma cell percentage ≥60%
  * Involved/un-involved serum free light chain ratio ≥100 and involved free light chain >100 mg/L.

    * 1 focal lesion on magnetic resonance imaging study (lesion must be >5 mm) in size
* Creatinine Clearance ≥ 60 ml/min. CrCl can be measured or estimated using Cockcroft-Gault method, MDRD, or CKD-EPI formulae
* Age ≥ 18 years at the time of signing the informed consent documentation
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 Absolute neutrophil count (ANC) ≥ 1.0 K/uL, hemoglobin ≥ 8 g/dL, and platelet count ≥ 75 K/uL, unless if cytopenias are deemed to be due disease at discretion of clinical investigator. Transfusions and growth factors are permissible.
* Adequate hepatic function, with bilirubin < 1.5 x the ULN, and AST and ALT < 3.0 x ULN.
* All study participants must be able to tolerate one of the following thromboprophylactic strategies: aspirin, low molecular weight heparin or warfarin (coumadin) or alternative anti-coagulant.
* All study participants must be registered into the mandatory eREMS® program, and be willing and able to comply with the requirements of REMS®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

* Patients receiving >1 cycle of prior treatment or concurrent systemic treatment for multiple myeloma

  * Treatment of hypercalcemia or spinal cord compression or aggressively progressing myeloma with current or prior corticosteroids is permitted
  * Bisphosphonates are permitted
  * Concurrent or prior treatment with corticosteroids for indications other than multiple myeloma is permitted
  * Prior treatment with radiotherapy is permitted
  * Prior treatment for smoldering myeloma is permitted with a washout period of 2 weeks from last dose. Smoldering patients previously treated with carfilzomib are excluded.
  * Patients with measurable disease who received up to one cycle of any therapy within 60 days with a washout period of 2 weeks from last dose (on a trial or outside a trial) are eligible
* Plasma cell leukemia
* POEMS syndrome
* Amyloidosis
* Has known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal (note that FEV1 testing is required for subjects suspected of having chronic obstructive pulmonary disease and subjects must be excluded if FEV1 <50% of predicted normal).
* Pregnant or lactating females. Because there is a potential risk for adverse events nursing infants secondary to treatment of the mother with carfilzomib in combination with lenalidomide. These potential risks may also apply to other agents used in this study.
* Uncontrolled hypertension or diabetes
* Active hepatitis B or C infection
* Subject is:

  * Seropositive for human immunodeficiency virus (HIV)
  * Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.*
  * Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
* Has significant cardiovascular disease with NYHA Class III or IV symptoms, EF<40% or hypertrophic cardiomyopathy, or restrictive cardiomyopathy, or myocardial infarction within 6 months prior to enrollment, or unstable angina, or unstable arrhythmia as determined by history and physical examination. Echocardiogram will be performed during screening evaluation.
* Pulmonary hypertension
* Has refractory GI disease with refractory nausea/vomiting, inflammatory bowel disease, or bowel resection that would prevent absorption of oral agents
* Uncontrolled intercurrent illness including but not limited to active infection or psychiatric illness/social situations that would compromise compliance with study requirements
* Significant neuropathy ≥Grade 3 or Grade 2 neuropathy with pain at baseline
* Contraindication to any concomitant medication, including antivirals or anticoagulation.
* Major surgery within 3 weeks prior to first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
assess the rate of MRD negativity | 2 years
  Patients with ≤ PR after completing 4 cycles will be included in the analysis of the primary objective and will be considered MRD positive. Patients who receive any study drug and have at least one post-baseline disease assessment will be considered evaluable for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Korde, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Maura F, Boyle EM, Coffey D, Maclachlan K, Gagler D, Diamond B, Ghamlouch H, Blaney P, Ziccheddu B, Cirrincione A, Chojnacka M, Wang Y, Siegel A, Hoffman JE, Kazandjian D, Hassoun H, Guzman E, Mailankody S, Shah UA, Tan C, Hultcrantz M, Scordo M, Shah GL, Landau H, Chung DJ, Giralt S, Zhang Y, Arbini A, Gao Q, Roshal M, Dogan A, Lesokhin AM, Davies FE, Usmani SZ, Korde N, Morgan GJ, Landgren O. Genomic and immune signatures predict clinical outcome in newly diagnosed multiple myeloma treated with immunotherapy regimens. Nat Cancer. 2023 Dec;4(12):1660-1674. doi: 10.1038/s43018-023-00657-1. Epub 2023 Nov 9. PMID 37945755
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm